CLINICAL TRIAL: NCT02568306
Title: A First Human Dose Trial Investigating Safety, Tolerability and Pharmacokinetics for Single Doses and Multiple Doses of NNC0165-1562 in Overweight to Obese But Otherwise Healthy Subjects.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: NN9747-4194; U1111-1164-6546 (Other: WHO)
Record Dates: First submitted 2015-10-02; First posted 2015-10-05 (Estimated); Last update posted 2018-07-13 (Actual); Status verified 2018-07

CONDITIONS: Metabolism and Nutrition Disorder; Obesity
MeSH Terms: conditions — Nutrition Disorders; Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- NNC0165-1562 (Experimental)
  Interventions: Drug: NNC0165-1562
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: NNC0165-1562 — Administered subcutaneously (s.c., under the skin) single dose [SD] or multiple dose [MD] with daily dosing.
  Arms: NNC0165-1562
Drug: placebo — Administered subcutaneously (s.c., under the skin) single dose [SD]) or multiple dose [MD] with daily dosing.
  Arms: Placebo

SUMMARY:
This trial is conducted in the United States of America. The aim of the trial is to investigate safety, tolerability and pharmacokinetics (the exposure of the trial drug in the body) for single doses and multiple doses of NNC0165-1562 in overweight to obese but otherwise healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Part I (SD):
* Male, aged 18-55 years (both inclusive) at the time of signing informed consent
* Body mass index (BMI) between 25.0 and 34.9 kg/m^2 (both inclusive). Overweight should be due to excess of adipose tissue, as judged by the investigator
* Considered to be generally healthy based on the medical history, physical examination, and the results of vital signs, electrocardiogram (ECG) and clinical laboratory tests performed during the screening visit, as judged by the investigator
* Part II (MD):
* Male or female, aged 18-55 years (both inclusive) at the time of signing informed consent
* Body mass index (BMI) between 27.0 and 39.9 kg/m^2 (both inclusive). Overweight should be due to excess of adipose tissue, as judged by the investigator
* Considered to be generally healthy based on the medical history, physical examination, and the results of vital signs, electrocardiogram (ECG) and clinical laboratory tests performed during the screening visit, as judged by the investigator

Exclusion Criteria:

* Any clinically significant weight change (at least 5% self-reported change during the previous 3 months), dieting attempts (e.g. participation in an organised weight reduction programme within the last 3 months), prior obesity surgery, or medications affecting body weight within 3 months prior to screening
* Male subjects who are not surgically sterilised (vasectomy) and are sexually active with female partner(s) who are not using a highly effective method of contraception (such as condom with spermicide) combined with a highly effective method of contraception for their non-pregnant female partner(s) (Pearl Index 1%, such as implants, injectables, oral contraceptives, intrauterine devices, diaphragm or cervical cap+spermicide), and/or intend to donate sperm in the period from screening until 3 months following administration of the investigational medical product
* Female subjects who are of child bearing potential (pre-menopausal and not surgically sterilised) and are sexually active with male partner(s) who are not surgically sterilised (vasectomy) and are not using highly effective contraceptive methods (Pearl Index 1%,such as implants, injectables, oral contraceptives, intrauterine devices, diaphragm or cervical cap+spermicide) combined with a highly effective method of contraception for their male partner(s) (e.g. condom with spermicide), and/or are pregnant, breast-feeding or intend to become pregnant) (applicable to Part II (MD) only)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 93 (Actual)
Dates: Start 2015-10-05 (Actual); Primary Completion 2017-02-07 (Actual); Study Completion 2017-02-07 (Actual)

PRIMARY OUTCOMES:
Number of treatment emergent adverse events (TEAEs), Part I (SD) | From time of dosing (Day1) until completion of the follow-up visit (Day 29)
Number of TEAEs, Part II (MD) | From time of dosing (Day 1) until completion of the follow-up visit (Day 85)

SECONDARY OUTCOMES:
The area under the NNC0165-1562 plasma concentration-time curve, Part I (SD) | From time 0 to 24 hours after a single s.c. dose. From baseline (Day 1) until the follow-up visit (Day 29)
The maximum plasma concentration of NNC0165-1562 after a single s.c. dose, Part I (SD) | From baseline (Day 1) until the follow-up visit (Day 29)
The time to maximum plasma concentration of NNC0165-1562 after a single s.c.dose, Part I (SD) | From baseline (Day 1) until the follow-up visit (Day 29)
The area under the NNC0165-1562 plasma concentration-time curve, Part II (MD) | From time 0 to 24 hours at steady state. From baseline (Day 1) until the follow-up visit (Day 85)
The maximum plasma concentration of NNC0165-1562 at steady state, Part II (MD) | From baseline (Day 1) until the follow-up visit (Day 85)
The time to maximum plasma concentration of NNC0165-1562 at steady state, Part II (MD) | From baseline (Day 1) until the follow-up visit (Day 85)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Tempe, Arizona, United States

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com